CLINICAL TRIAL: NCT04914806
Title: Association Between Premature Birth and Its Comorbidities With NO and the HPG Activation at Minipuberty
Brief Title: Infantile NO Replenishment as a New Therapeutic Possibility
Acronym: miniNO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: URI-NKUA (Unknown); University Hospital, Lille (Other); Centre Hospitalier Universitaire Vaudois (Other); European Commission (Other)
Responsible Party: Principal Investigator, Soultana (Tania) Siahanidou, Professor, National and Kapodistrian University of Athens
Other Study IDs: miniNO
Record Dates: First submitted 2021-05-27; First posted 2021-06-07 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Prematurity; Respiratory Distress Syndrome, Newborn
Keywords: preterm birth; neurodevelopment; cardiometabolic; minipuberty
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for hormones and metabolic parameters; genetic and epigenetic screening for NO pathway.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Infants treated with iNO (from birth to 1-3 weeks of life) or sequential treatment with iNO and sildenafil (for 1 to 3 months).
- Controls: Infants matched to cases (gestational/postnatal age, gender, disease state) and no iNO treatment.

SUMMARY:
Case-control study of inhaled Nitric Oxide (iNO) treatment of full-term and preterm infants. The main objective of this study is to investigate the association between premature birth and its later comorbidities (neuroendocrine, metabolic, cognitive, etc) with iNO treatment and the maturation of the HPG axis during minipuberty.

DETAILED DESCRIPTION:
In preterm infants, inhaled NO (iNO) is routinely used to treat respiratory failure and pulmonary hypertension, while preclinical studies have shown that it markedly increases NO concentrations in the brain. Animal and human studies have shown that NO deficiency may jeopardize the establishment of a mature and functional HPG axis whereas it is also associated with a series of comorbidities affecting the overall brain development (e.g. sensory, fertility and cognitive functions). Prematurity has been associated with a series of non-communicable diseases of major importance in public health, including neurodevelopmental impairments, metabolic abnormalities (e.g. obesity, type 2 diabetes mellitus, impaired glucose tolerance) and cardiovascular disease. This study aims to evaluate the associations between altered minipuberty in preterm infants and the later development of multi-comorbidities (mental and non-mental disorders), and identify the possible implication of the NO pathway as a causative mechanism.

Specific objectives :

1. Assess the efficiency of NO replenishment therapy (i.e. role of NO pathway) as a therapeutic against alterations of minipuberty resulting from preterm birth.
2. Assess the efficiency of NO replenishment therapy (i.e. role of NO pathway) as a therapeutic against the multi-comorbidities (mental and non-mental disorders) related to altered minipuberty as a result of preterm birth.

ELIGIBILITY:
Inclusion Criteria:

* Preterm (GA<37 weeks) or full-term (≥37 weeks of gestation) infants
* Requiring respiratory support
* Admitted to Neonatal Care Unit

Exclusion Criteria:

* Severe congenital anomalies
* Suspected major chromosomal anomalies
* Infants judged by the physician as nonviable

Ages: 1 Day to 3 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm and full-term infants admitted to the Neonatal Unit due to respiratory distress.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gonadotrophin levels | up to 9 months of age
  Serial blood levels of gonadotrophins (FSH and LH)
Body fat and fat-free mass | up to 9 months of age
  Serial fat and fat-free mass measurements by air displacement plethysmography
HOMA-IR | up to 9 months
  Serial measurements of blood glucose/insulin (HOMA-IR)
Bayleys scale score | at 9 months of age
  The Bayley Scales of Infant and Toddler Development will be used to assess neurodevelopment. Values <85 indicate developmental delay.

SECONDARY OUTCOMES:
Otoacoustic emissions | up to 9 months
  Serial otoacoustic emissions as a screening test for hearing ability
Fundoscopy | up to 9 months
  Ophthalmological follow-up for retina and visual assessment
gusto-facial reflex | at 3 and 9 months of age
  Assessment of olfaction will be performed using a citrus, vanilla or neutral odor, delivered on a cotton swab. The facial expressions in reaction to the different smells (the gusto-facial reflex) will be monitored while at rest (baseline), and in response to stimuli.
Leptin levels | up to 9 months
  Serial measurements of serum leptin levels

CONTACTS AND LOCATIONS:
Overall Officials: George P. Chrousos, Professor, Study Chair — URI-NKUA, Athens, Greece, 11527
Locations (3):
- Centre Hospitalier Regional Et Universitaire de Lille, Lille, France
- URI-NKUA, Athens, Greece
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided